CLINICAL TRIAL: NCT06902298
Title: Personalized Ultrasonic Brain Stimulation for Depression: A Study of Target Engagement and Mood Effects
Brief Title: Personalized Ultrasonic Brain Stimulation for Depression (R61)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Brian Mickey (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor-Investigator, Brian Mickey, Professor, University of Utah
Organization: University of Utah (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB_00148802R61; R61MH134943 (NIH)
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-03

CONDITIONS: Major Depressive Episode; Depression - Major Depressive Disorder; Treatment-Resistant Major Depressive Disorder
Keywords: ultrasonic neuromodulation; low-intensity focused ultrasound

STUDY DESIGN:
Intervention Model Description: Two brain targets will be stimulated sequentially. The order of the two targets will be randomized.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: All individuals are masked except the device operator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Group 1: SCC-ALIC (Experimental): Low-intensity transcranial focused ultrasound stimulation (LTFUS) is delivered to the subgenual cingulate cortex (SCC) at the first stimulation visit, then LTFUS is delivered to the anterior limb of the internal capsule (ALIC) at the second stimulation visit.
  Interventions: Device: LTFUS to SCC; Device: LTFUS to ALIC
- Group 2: ALIC-SCC (Experimental): Low-intensity transcranial focused ultrasound stimulation (LTFUS) is delivered to the anterior limb of the internal capsule (ALIC) at the first stimulation visit, then LTFUS is delivered to the subgenual cingulate cortex (SCC) at the second stimulation visit.
  Interventions: Device: LTFUS to SCC; Device: LTFUS to ALIC

INTERVENTIONS:
Device: LTFUS to SCC — Low-intensity transcranial focused ultrasound delivered to subgenual cingulate cortex
Device: LTFUS to ALIC — Low-intensity transcranial focused ultrasound delivered to anterior limb of internal capsule

SUMMARY:
This study will evaluate a new form of non-invasive brain stimulation for individuals with depression. Personalized low-intensity transcranial focused ultrasound stimulation will be delivered using a range of stimulation parameters during psychological and physiological monitoring. Individualized optimal targets will be selected using structural MRI and diffusion tractography. Brain target engagement will be evaluated using functional MRI.

DETAILED DESCRIPTION:
This R61 project has 3 aims:

1. To determine whether stimulation engages the subcallosal cingulate (SCC) in an intensity-dependent manner
2. To examine the degree of specificity of neuromodulation by contrasting the neural effects of stimulating two spatially distinct targets versus sham
3. To evaluate safety, tolerability, and side effects

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65, any gender.
2. Primary diagnosis of DMS-5 major depressive disorder (MINI).
3. Current moderate-to-severe depressive episode, without psychotic features, lasting at least 2 months (MINI).
4. Self-rated 16-item Quick Inventory of Depressive Symptomatology (QIDS) total score > 10.
5. History of at least 2 failed trials of evidence-based antidepressant medication and/or psychotherapy (at least one trial during the current depressive episode).
6. Stated willingness to comply with all study procedures and avoid changes to psychiatric treatments (medications, psychotherapy) for the duration of the study.
7. For participants of reproductive potential: negative pregnancy test or use of highly effective contraception for at least 1 month prior to baseline; agreement to use such a method throughout the study.
8. Capacity to provide informed consent; provision of a signed and dated consent form
9. Currently are under the care of a licensed psychiatrist or other mental health care provider, or a licensed addiction medicine specialist and agrees to promptly inform the investigator or the study staff of any change in these providers.
10. Agrees to allow any and all forms of communication between the investigators/study staff and any healthcare provider who currently provides and/or has provided service to the patient/subject within at least two years of study enrollment for the purposes of eligibility confirmation or in case of a safety event.
11. Agrees to provide the name and verifiable contact information (email and mailing addresses, mobile and land-line phone numbers, as applicable) of at least two persons 22 years or older who reside within a 60-minute drive of the patient's residence. Subject agrees that in the event of a safety concern or event during study participation, research staff is at liberty to contact these individuals if the subject does not respond to contact attempts.

Exclusion Criteria:

1. History of serious brain injury or other neurologic disorder.
2. Poorly managed general medical condition.
3. Pregnant or breast feeding.
4. Implanted device in the head or neck.
5. MRI intolerance or contraindication.
6. Brain stimulation treatment such as ECT, TMS, or VNS (past month).
7. Recent change in antidepressant treatments (past month).
8. 8. Moderate-High Risk of Suicide according to the Columbia - Suicide Severity Rating Scale (C-SSRS) Screen Version - Recent (answers YES to Question 3 and NO to Question 6 (Moderate risk) or YES to Question 4, 5, or 6 (High risk)) and/or in the clinical judgement of the PI or a study psychiatrist
9. Suicidal behavior (past year).
10. Serious suicide attempt 33 (lifetime).
11. Moderate-to-severe substance use disorder (MINI, past 3 months).
12. Obsessive compulsive disorder, primary diagnosis (MINI, past month).
13. Posttraumatic stress disorder, primary diagnosis (MINI, past month).
14. Bipolar-spectrum disorder (MINI, lifetime).
15. Schizophrenia-spectrum disorder (MINI, lifetime).
16. Neurocognitive disorder (DSM-5, past year).
17. Severe personality disorder.
18. Clinically inappropriate for participation in the study as determined by the study team.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Modulation of SCC activity during SCC stimulation | Days 14, 21, 28
  Functional MRI is used to quantify modulation of SCC activity during SCC stimulation
Modulation of SCC activity during ALIC stimulation | Days 14, 21
  Functional MRI is used to quantify modulation of SCC activity during ALIC stimulation
Study dropout | From enrollment to the end of participation at 7 weeks
  Dropout or withdrawal due to stimulation-related adverse effects

SECONDARY OUTCOMES:
PANAS-X | Immediately before and after each LTFUS on Days 14, 21, 28
  Positive and Negative Affect Schedule, Expanded Form
MADRS | Days 14, 21, 28, 35, 49
  Montgomery-Asberg Depression Rating Scale
HDRS-6 | Days 0, 14, 15, 21, 22, 28, 29, 35, 49
  6-item Hamilton Depression Rating Scale
IDS-SR | Days 0, 14, 21, 28, 35, 49
  Inventory of Depressive Symptomatology, Self-Rated
GAD-7 | Days 0, 14, 21, 28, 35, 49
  7-item Generalized Anxiety Disorder Scale
YMRS | Days 0, 14, 15, 21, 22, 28, 29, 35, 49
  Young Mania Rating Scale
C-SSRS | Days 0, 14, 15, 21, 22, 28, 29, 35, 49
  Columbia Suicide Severity Rating Scale, Screen Version
GASE | Days 15, 22, 29
  Generic Assessment of Side Effects scale
MoCA | Days 14, 15, 49
  Montreal Cognitive Assessment

CONTACTS AND LOCATIONS:
Overall Officials: Brian J Mickey, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided